CLINICAL TRIAL: NCT04015089
Title: Randomized, Parallel, Double-blind Study With a Partially Hydrolyzed Infant Formula With Cow's Milk Protein vs a Formula With Intact Protein to Assess Growth and Impact on the Gastrointestinal Manifestations of Colic in the Healthy Infant.
Brief Title: Infant Formula With Partially Hydrolyzed Cow's Milk Protein Versus a Formula With Intact Protein
Acronym: VEGY-UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratorios Ordesa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EC-MAGICO-01-18; MAGICO (Other: Ordesa)
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Infant Colic
Keywords: Infant formula; Partially hydrolized protein infant formula
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially hydrolyzed formula (pHF) (Experimental): Infants fed exclusively with a infant formula based on partially hydrolyzed serum cow's milk proteins.
  Interventions: Dietary Supplement: Partially hydrolyzed formula (pHF)
- Standard formula (SF) (Active Comparator): Infants fed exclusively with a standard formula based on intact cow's milk proteins
  Interventions: Dietary Supplement: Standard formula (SF)

INTERVENTIONS:
Dietary Supplement: Partially hydrolyzed formula (pHF) — Infant formula with partially hydrolyzed protein
  Arms: Partially hydrolyzed formula (pHF)
Dietary Supplement: Standard formula (SF) — Infant formula with intact protein
  Arms: Standard formula (SF)

SUMMARY:
Randomized, parallel, double-blind clinical trial, comparing a partially hydrolyzed serum proteins infant formula with a conventional formula with intact protein in healthy infants that suffer from colic

DETAILED DESCRIPTION:
Demonstrate that an infant formula with partially hydrolized cow's milk protein of serum proteins is equivalent to an intact protein formula in healthy children in terms of safety of use and suitability, to prove that it can be a alternative with digestive health benefits in healthy children with infant colic.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as nursing colic according to Roma IV criteria.
* Infants who have received breastfeeding at least 2 weeks.
* Infants who at the time of inclusion in the study whose parents/legal guardians voluntarily decide not to continue exclusive breastfeeding or only maintain it in residual form (less than 20% of the daily intake, one breast intake per day).
* Full-term infants (>37 weeks of gestation).
* Infants with weight suitable for their gestational age (2500-4500g).
* Normal APGAR score: 7-10.
* Infants between 2 and 8 weeks of life.
* Infants whose parents/legal guardians have signed informed consent.
* Infants with good availability of clinical follow-up until the end of the study.

Exclusion Criteria:

* Infants fed from birth with exclusive infant formula.
* Infants with congenital diseases or malformations that may affect growth.
* Infants with major medical conditions that require chronic medication or close medical checks.
* Infants who have taken any type of antibiotics or probiotics prior to the study.

Ages: 2 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2018-07-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Growth standard calculated z-scores | From baseline to 3 months after starting with the formula
  Using Z-scores including: weight (g), size (cm) and cranial perimeter (cm)
Symptoms associated with infant colic | From baseline to 3 months after starting with the formula
  Hours of crying, wakefulness, sleep for 24 hours, by adapting Barr's crying letter

SECONDARY OUTCOMES:
Growth standard calculated z-scores | At 6, 9 and 12 months old.
  Using Z-scores including: weight (g), size (cm) and cranial perimeter (cm)
Gatrointestinal tolerance recording | Baseline, 1, 2 and 3 months follow-up visit, and 6, 9 months old
  Record in the patient's diary stool patterns (depositional rhythm and quality of faeces)
Infant illness and infection outcomes | Baseline, 1, 2 and 3 months follow-up visit, and 6, 9 months old
  Specific parent-reported infant symptoms (digestive, respiratory or other infections)
Behaviour/temperament test | 1, 6, 12 months old
  Infant Behavior Questionnaire-Revised test: For this study, the very short form validated in Spanish that includes 37 items will be applied. Parents are asked to rate the frequency of specific, temperament-related behaviors observed during the last week.
Assessment of supplementary food | At 6 and 9 months old
  Investigator will collect data from the timetable for introduction of the different food groups
Food survey at the first year of life | At 12 months old
  Investigator will conduct a food consumption frequency survey
Product safety | At 1, 2 and 3 months follow-up visit, and 6, 9 months old
  Assessment of acceptance of the formula and record of potential adverse or side effects related to taking the product.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Martin Martínez, Principal Investigator — Consorci Sanitari de Terrassa; Gemma Colomé Rivero, Principal Investigator — Fundació Hospital de Nens de Barcelona
Locations (2):
- Spain (2):
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Fundació Hospital de Nens, Barcelona